CLINICAL TRIAL: NCT05597657
Title: Normal Variation of T1 Values With Cardiac Magnetic Resonance in Healthy Individuals
Acronym: NATIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cardiovascular Academy (DCA) (Unknown); Eva og Henry Frænkels Mindefond (Other); Snedkermester Sophus Jacobsen and hustru Astrid Jacobsens Foundation (Other)
Responsible Party: Principal Investigator, Katrine Aagaard Myhr, Principital Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-21025256
Record Dates: First submitted 2022-05-25; First posted 2022-10-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Magnetic Resonance; T1 Mapping; Healthy Individuals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluid administration (substudy 2) (Other)
  Interventions: Other: Fluid administration (Fresenius Kabi Sodium Chloride 0.9%)

INTERVENTIONS:
Other: Fluid administration (Fresenius Kabi Sodium Chloride 0.9%) — All participants in substudy 2 will be administered 2 liters of isotonic saline infusion (Fresenius Kabi Sodium Chloride 0.9%) intravenously. CMR and echocardiography will be performed before and after infusion.

SUMMARY:
The purpose of the study is to determine the normal variation of T1 values with cardiac magnetic resonance in healthy individuals with respect to reproducibility, changes over time, and dependency on hydration status.

DETAILED DESCRIPTION:
T1 mapping with cardiac magnetic resonance (CMR) is a novel non-invasive technique to quantitatively characterize the myocardium. T1 mapping is a surrogate marker of myocardial edema and fibrosis, and has the potential to be implemented in the diagnosis and follow-up of various cardiac diseases. However, there is limited data on the natural variation of T1 mapping in healthy individuals.

The study comprises three substudies:

1. Reproducibility: Two identical CMR examinations with T1 mapping will be performed on the same day .
2. Hydration changes: Participants will receive two liters of isotonic saline intravenously between two identical CMR with T1 mapping and echocardiographic examinations. The post-fluid order of CMR and echocardiography will be randomized.
3. Time changes: Participants will undergo CMR with T1 mapping at baseline, at 6-months follow-up, and at 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89 years
* Healthy

Exclusion Criteria:

* Chronic disease (e.g. cardiovascular disease, rheumatological disease, lung disease)
* Medications affecting the cardiovascular system (e.g. antihypertensives, statins, anticoagulants)
* Contraindications for CMR (claustrophobia, pregnancy, magnetic metallic implants)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change in T1 values (substudy 1) | Through study completion, an average of 1 year
  Change in T1 values between two consecutive scans on the same day
Change of T1 values (substudy 2) | Through study completion, an average of 1 year
  Change in T1 values after fluid administration
Change in T1 values (substudy 3) | Through study completion, an average of 1 year
  Change in T1 values over time (baseline, 6 months, 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Katrine A Myhr, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data can be provided upon request
Time Frame: From study end
Access Criteria: Researchers who provide a methodological sound proposal